CLINICAL TRIAL: NCT07189273
Title: Eye Medication Administration Experiences of Parents of Children Aged 2-6 Years Who Underwent Strabismus Surgery: A Qualitative Study
Brief Title: Parents' Experiences of Administration Eye Drops
Status: Completed | Type: Observational
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Yeliz Sapulu Alakan, Ph.D., Uludag University
Other Study IDs: Strabismus Surgery
Record Dates: First submitted 2025-09-09; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Strabismus; Strabismus Surgery
Keywords: child; Strabismus surgery; Eye drop administration; Caregiver
MeSH Terms: conditions — Strabismus

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to determine the experiences of parents of children aged 2-6 years who underwent strabismus surgery in eye drop administration and the cooperation of their children.

Methods: This semi-structured qualitative study was conducted with caregivers (n=13) of children aged 2-6 years who underwent strabismus surgery at the eye clinic of a university hospital in a province in the northwest of X. Data were collected through phone interviews held with children's parents on the third postoperative day. The interviews were audio-recorded, and the content of the recordings was analyzed using traditional content analysis.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children aged 2-6 years
* Children who had never undergone eye surgery before
* Children who had strabismus surgery for the first time

Exclusion Criteria:

* Parents of children with physical and mental developmental retardation
* Parents with cognitive disorders
* Parents with hearing disorders

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Parents of children aged 2-6 years who had never undergone eye surgery before and had strabismus surgery for the first time were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2024-04-05 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-07-21 (Actual)

PRIMARY OUTCOMES:
Data collection form | Data was collected on the third day after the children were discharged.
  Development of Data Collection Form: A data collection form was developed by researchers based on the relevant literature. The form consisted of two sections.
  Section I: This section consisted of eight descriptive questions regarding the sociodemographic characteristics of children and their parents.
  Section II: This section consisted of seven semi-structured questions to evaluate the experiences of parents of children aged 2-6 years who underwent strabismus surgery when administering eye drops to their children, as well as the children's cooperation. The total number of questions in the form was 15.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludag University, Bursa, Nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
As this is a qualitative study, all data will be included in the article.

REFERENCES:
- [Background] Hirji N, Jones S, Thompson G. The causes of distress in Paediatric outpatients receiving dilating drops. Open J Ophthalmol. 2012;2:21.